CLINICAL TRIAL: NCT00937144
Title: Endothelial Function in Patients With Sickle Cell Anemia Before and After Sildenafil
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: we didnt recieved the medicine
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: baruch padeh poria medical center, ministry of health, Israel
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SCA123-CTIL
Record Dates: First submitted 2008-09-24; First posted 2009-07-10 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2009-07

CONDITIONS: Sickle Cell Anemia
Keywords: endothelial function; endothelial progenitor stem cells
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- viagra (Experimental): viagra versus placebo will be given to patients with sickle cell anemia
  Interventions: Drug: Viagra (Sildenafil)
- placebo (Placebo Comparator): viagra versus placebo will be given to patients with sickle cell anemia
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Viagra (Sildenafil) — Viagra treatment to patients with sickle cell anemia.
  Arms: viagra
Drug: placebo
  Arms: placebo

SUMMARY:
The investigators would like to study the endothelial function in sickle cell patients without pulmonary hypertension in an in vivo method during a steady state condition before and after sildenafil treatment for 1 month, and to study the effects of this nitric oxide donor by measuring the Flow Mediated Dilatation, by measuring endothelial progenitor stem cells colonies, and by measuring the effect of therapy on markers of inflammation (cell adhesion molecules and cytokines).

ELIGIBILITY:
Inclusion Criteria:

* patients with sickle cell anemia

Exclusion Criteria:

* patients with sickle cell anemia during acute crisis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-09; Primary Completion 2009-09 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
endothelial function before and after viagra treatment to patients with sickle cell anemia without pulmonary hypertension | January 2009 till January 2011

CONTACTS AND LOCATIONS:
Locations (1):
- Baruch Padeh Poria Medical Center, Tiberias, Lower Galilee, Israel